CLINICAL TRIAL: NCT02663401
Title: Impact of a Front-of-pack Nutrition Label on the Nutritional Quality of Purchases in Campus Cafeterias
Acronym: 5-C CROUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Paris 13 (Other)
Responsible Party: Principal Investigator, Serge HERCBERG, Professeur des Universités - Praticien Hospitalier, University of Paris 13
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CROUS_NICE
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Food Labelling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control situation in campus cafeterias where no labelling of food is proposed
- Front-of-pack labelling (5-CNL) (Experimental): Introduction of the 5-CNL front-of-pack nutrition label on shelf display tags for every food and beverage sold in the campus cafeteria. Communication campaigns accompanying the introduction of the label
  Interventions: Behavioral: Front-of-pack labelling 5-CNL

INTERVENTIONS:
Behavioral: Front-of-pack labelling 5-CNL — Introduction of the 5-CNL Front-of-pack nutrition label on shelf display tags for every food and beverage sold in the cafeteria
  Arms: Front-of-pack labelling (5-CNL)

SUMMARY:
This study evaluates the impact of the introduction of a front-of-pack nutrition label on fods and beverages sold in a campus cafeteria in France on the nutritional quality of purchases. The design involves one site with the intervention and one control site with the same consumer and product characteristics.

DETAILED DESCRIPTION:
The introduction of front-of-pack nutrition labelling is thought to help consumers making healthier choices at the point of purchase.

Recently, the French government is considering the introduction of the 5-Colour Nutrition Label as a front-of-pack nutrition label.

Evaluations of the 5-CNL suggest it is efficient in helping consumers making healthier choices. However, its impact in vulnerable populations has not yet been tested.

Students are thought to be a vulnerable population due to their limited resources and to their unhealthy food choices.

The objective of the present study is to investigate the impact of the introduction of the 5-CNL in campus cafeterias on the nutritional quality of food purchases.

The intervention is conducted during several months, with another similar cafeteria serving as control for the intervention.

Data on purchases is collected regularly, and the nutritional quality of purchases is evaluated over time between the intervention situation and the control situation

ELIGIBILITY:
Inclusion Criteria:

* All subjects purchasing foods or beverages in the selected campus cafeterias

Exclusion Criteria:

* None

No individual data is collected. Only purchases data is collected (cash register sales data)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Overall nutritional quality of purchases | Every 15 days, up to 6 months
  Overall nutritional quality of purchases evaluated using the Food Standard Agency nutrient profiling system

SECONDARY OUTCOMES:
Energy content of purchases | Every 15 days, up to 6 months
  Energy content of the purchases (kcal/100g)
Saturated fat content of purchases | Every 15 days, up to 6 months
  saturated fat content of the purchases (g/100g)
Sugar content of purchases | Every 15 days, up to 6 months
  Sugar content of the purchases (g/100g)
Sodium content of purchases | Every 15 days, up to 6 months
  Sodium content of the purchases (mg/100g)
Fibers content of purchases | Every 15 days, up to 6 months
  Fiber content of the purchases (g/100g)
Protein content of purchases | Every 15 days, up to 6 months
  Protein content of the purchases (g/100g)

CONTACTS AND LOCATIONS:
Locations (1):
- CROUS Nice - Toulon, Nice, France

IPD SHARING:
Plan to Share IPD: No